CLINICAL TRIAL: NCT04089098
Title: Characterizing VOLume and Vasopressor Therapy in Patients With Hemodynamic instAbility (VOLTA)
Brief Title: VOLume and Vasopressor Therapy in Patients With Hemodynamic instAbility
Acronym: VOLTA
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Sirak Petros, MD, Professor, University of Leipzig
Other Study IDs: VOLTA-01
Record Dates: First submitted 2019-09-03; First posted 2019-09-13 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hemodynamic Instability; Shock; Septic Shock
Keywords: fluid resuscitation; shock; volume challenge; passive leg raising; renal perfusion; fluid responsiveness
MeSH Terms: conditions — Shock; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — norepinephrine renin copeptin A cortisol angiopoietin-2 cystatin C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: passive leg raising versus mini volume challenge — Blood samples will be collected and ultrasound evaluation of renal perfusion conducted in study participants immediately before conducting passive leg raising (PLR). PLR will then be carried out on study participants, followed by MVC. PLR- and/or MVC-responsive patients will receive a further 700 ml fluid immediately after the MVC. Renal perfusion will be further assessed 1 and 24 hours after the MVC.

SUMMARY:
This prospective observational study will include critically ill patients with hemodynamic compromise. It will compare passive leg raising and a mini volume challenge (MVC) carried out on every patient sequentially. The endogenous release of stress hormones will also be assayed in order to investigate their modifying effect on the hemodynamic reaction of the participants. The effect of fluid resuscitation on renal perfusion will also be assessed and the data compared with the release of cystatin C.

DETAILED DESCRIPTION:
Fluids are administered either before starting with or during ongoing vasopressor treatment in critically ill patients with hemodynamic instability. The endogenous release of stress hormones, namely renin, vasopressin, norepinephrine and cortisol, may be variable in critically ill patients, which may have a modifying effect on the hemodynamic response. Passive leg raising (PLR), a validated, simple and dynamic test, is currently recommended for testing fluid responsiveness. The test might possibly be false negative under extreme dehydration or increased intra-abdominal pressure. This prospective observational study aims to compare PLR and MVC with 300 ml Ringer acetate solution administered as a bolus within 5 minutes in critically ill medical patients with a hemodynamic instability. MVC will be carried out in every participant following PLR. Blood samples will be collected immediately before PLR for measurement of renin, copeptin A, cortisol and norepinephrine in those patients not yet receiving a vasopressor. These biomarkers will be compared with the Magnitude of fluid responsiveness. Additionally, renal resistive index will be assessed with ultrasound immediately before PLR and 1 and 24 hours after fluid challenge and the data compared with Initial serum cystatin C in those patients who have not yet developed acute renal failure. Blood samples for measurement of angiopoietin-2, a marker of capillary leak, will be drawn immediately before PLR and the data will be correlated with the amount of fluid required for Initial resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* mean arterial pressure <65 mm Hg and/or
* blood lactate >2 mmol/l and/or
* mottling or capillary refill >3 seconds and/or
* oliguria and
* critical care decision for testing fluid responsiveness

Exclusion Criteria:

* cardiopulmonary resuscitation
* uncontrolled bleeding
* irreversible brain damage
* pregnancy and lactation
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill adult medical patients with signs of hemodynamic instability
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in blood pressure under PLR vs. MVC | immediately at the end of the MVC
  changes in mean arterial pressure with PLR vs. MVC

SECONDARY OUTCOMES:
Hemodynamic changes with PLR vs. MVC | immediately at the end of the MVC
  Changes in cardiac Output under PLR vs. MVC
fluid requirement and endogenous stress response | at the end of the first 3 hours of fluid resuscitation
  correlation between fluid requirement and the level of endogenous renin, copeptin A, cortisol and norepinephrine
fluid administration versus renal perfusion | 1 and 24 hours after initial fluid resuscitation
  renal resistive index will be assessed 1 and 24 hours after the Initial fluid resuscitation
fluid administration and capillary leak | at the end of the first 3 hours of fluid resuscitation
  Fluid resuscitation in the first 3 hours vs. initial serum angiopoietin-2

CONTACTS AND LOCATIONS:
Overall Officials: Sirak Petros, MD, Study Director — University Hospital of Leipzig, Medical ICU
Locations (1):
- University Hospital of Leipzig, Leipzig, Saxony, Germany